CLINICAL TRIAL: NCT05480865
Title: A Phase 1 Study of the SHP2 Inhibitor BBP-398 (Formerly Known as IACS-15509) in Combination With the KRAS-G12C Inhibitor Sotorasib in Patients With Advanced Solid Tumors and a KRAS-G12C Mutation
Brief Title: SHP2 Inhibitor BBP-398 in Combination With Sotorasib in Patients With Advanced Solid Tumors and a KRAS-G12C Mutation
Acronym: Argonaut
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Navire Pharma Inc., a BridgeBio company (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NAV-1003
Record Dates: First submitted 2022-07-15; First posted 2022-07-29 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Solid Tumor, Adult; Metastatic Solid Tumor; Metastatic NSCLC; Non Small Cell Lung Cancer
Keywords: KRAS-G12C mutation; SHP2; MAPK-pathway alterations; NSCLC
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung | interventions — sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Dose Escalation: BBP-398 Level 1 and sotorasib (Experimental): BBP-398 dose Level 1 capsules administered once a day (QD) for a 28-day treatment cycle in combination with sotorasib tablets administered once a day (QD) for a 28-day treatment cycle
  Interventions: Drug: BBP-398; Drug: sotorasib
- Dose Escalation: BBP-398 Level 2 and sotorasib (Experimental): BBP-398 dose Level 2 capsules administered once a day (QD) for a 28-day treatment cycle in combination with sotorasib tablets administered once a day (QD) for a 28-day treatment cycle
  Interventions: Drug: BBP-398; Drug: sotorasib
- Dose Escalation: BBP-398 Level 3 and sotorasib (Experimental): BBP-398 dose Level 3 capsules administered once a day (QD) for a 28-day treatment cycle in combination with sotorasib tablets administered once a day (QD) for a 28-day treatment cycle
  Interventions: Drug: BBP-398; Drug: sotorasib
- Dose Expansion/Optimization: BBP-398 Dose Regimen 1 and sotorasib (Experimental): BBP-398 Dose Regimen 1 capsules administered once a day (QD) for a 28-day treatment cycle in combination with sotorasib tablets administered once a day (QD) for a 28-day treatment cycle
  Interventions: Drug: BBP-398; Drug: sotorasib
- Dose Expansion/Optimization: BBP-398 Dose Regimen 2 and sotorasib (Experimental): BBP-398 Dose Regimen 2 capsules administered once a day (QD) for a 28-day treatment cycle in combination with sotorasib tablets administered once a day (QD) for a 28-day treatment cycle
  Interventions: Drug: BBP-398; Drug: sotorasib

INTERVENTIONS:
Drug: BBP-398 — BBP-398 administered orally
Drug: sotorasib — sotorasib administered orally

SUMMARY:
This is a Phase 1 study of BBP-398, a SHP2 inhibitor, in combination with sotorasib, a KRAS-G12C inhibitor (KRAS-G12Ci), in patients with a KRAS-G12C mutation.

The study involves 2 parts: Phase 1a Dose Escalation and Phase 1b Dose Expansion/Optimization.

DETAILED DESCRIPTION:
The primary objectives for Phase 1a Dose Escalation are to evaluate safety and tolerability, and recommend a phase 1b dose (RP1bD) of the combination.

The primary objectives for Phase 1b Dose Expansion/Optimization are to evaluate safety and tolerability, and the antitumor activity (defined by the ORR assessed by the investigator according to RECIST v1.1) of BBP-398 when used in combination with sotorasib across two dose regimens in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) with a KRAS-G12C mutation and who are KRAS-G12Ci naïve, and recommend a phase 2 dose (RP2D) of the combination.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients must have histologically documented, locally advanced and unresectable, or metastatic solid tumor with documentation of a KRAS-G12C mutation within 2 years prior to screening.
* Patients must have measurable disease by RECIST v1.1.
* Patients must have a minimum life expectancy of >12 weeks after start of study treatment.
* Patients must have progression or disease recurrence on or after all available standard of care therapies.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
* Patients must have adequate organ function.

Key Exclusion Criteria:

* Patients that have participated in an interventional clinical study within the last 4 weeks.
* Patients that have received radiotherapy or proton therapy with a limited field of radiation for palliation within 1 week of the start of study treatment, OR radiation to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the start of study treatment.
* Patients with untreated and/or active CNS metastases.
* Patients that have a history of allogenic bone marrow transplant.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
Phase 1a Dose Escalation Primary Objective: Incidence and Severity of Treatment-Emergent Adverse Events, Serious Adverse Events, and Dose Limiting Toxicities | Completion of 1 Cycle (28 days)
  Number of patients experiencing treatment-emergent adverse events, serious adverse events, including changes in lab parameters, vital signs and electrocardiogram changes; duration, and severity based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Phase 1b Dose Expansion/Optimization Primary Objective: Incidence and Severity of Treatment-Emergent Adverse Events, and Serious Adverse Events | Completion of 1 Cycle (28 days)
  Number of patients experiencing treatment-emergent adverse events, serious adverse events, including changes in lab parameters, vital signs and electrocardiogram changes; duration, and severity based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Phase 1b Dose Expansion/Optimization Primary Objective: Overall Response Rate (ORR) | 8 weeks
  Complete Response (CR) + Partial Response (PR) rates, defined by RECIST v1.1

SECONDARY OUTCOMES:
Phase 1a Dose Escalation Secondary Objectives: Overall Response Rate (ORR) | 8 weeks
  Complete Response (CR) + Partial Response (PR) rates, defined by RECIST v1.1
Duration of response | 8 weeks
  Defined by RECIST v1.1
Progression Free Survival (PFS) | 8 weeks
  Time from treatment start to progression of disease or death by any cause
Overall survival (OS) | 8 weeks
  Time from treatment start to death
Maximum Observed Plasma Concentration (Cmax) of BBP-398 | Cycle 2 Day 1
  Maximum plasma concentration of BBP-398 in combination with sotorasib
Time to Cmax (Tmax) of BBP-398 | Cycle 2 Day 1
  Amount of time to reach Cmax of BBP-398 in combination with sotorasib
Area under the plasma concentration-time curve (AUC) of BBP-398 | Cycle 2 Day 1
  Area under the plasma concentration versus time curve of BBP-398 in combination with sotorasib
Half-life (T1/2) of BBP-398 | Cycle 2 Day 1
  Terminal half-life of BBP-398 in combination with sotorasib
Observed Maximum Plasma Concentration (Cmax) of sotorasib | Cycle 2 Day 1
  Maximum plasma concentration of sotorasib in combination with BBP-398
Time to Cmax (Tmax) of sotorasib | Cycle 2 Day 1
  Amount of time to reach Cmax of sotorasib in combination with BBP-398
Area under the plasma concentration-time curve (AUC) over dosing interval of sotorasib | Cycle 2 Day 1
  Area under the plasma concentration versus time curve of sotorasib in combination with BBP-398
Half-life (T1/2) of sotorasib | Cycle 2 Day 1
  Terminal half-life of sotorasib in combination with BBP-398
Circulating and intratumoral target engagement biomarkers of BBP-398 activity in combination with sotorasib | 24 months
  Raw, normalized, and/or baseline adjusted analyte signal

CONTACTS AND LOCATIONS:
Locations (25):
- Australia (6):
  - Cancer Research SA, Adelaide, South Australia
  - Southern Oncology Clinical Research Unit, Adelaide, South Australia
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria
  - One Clinical Research, Perth, Western Australia
  - St John of God Subiaco Hospital, Subiaco, Western Australia
  - Orange Health Service, Orange
- Rigshospitalet, Copenhagen, Denmark
- France (5):
  - Institute Bergonie, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - CHU Grenobles Aples, Grenoble
  - Hopital Bichat-Claude Bernard, Paris
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
- St. Luke's Hospital S.A., Thessaloniki, Greece
- Italy (4):
  - Careggi University Hospital, Florence, Largo Brambilla
  - Spedali Civili - Brescia, Brescia
  - Istituto Nazionale Tumori (INT) "Fondazione G. Pascale", Napoli
  - U.O.C Oncoematologia AOU "Luigi Vanvitelli", Napoli
- Netherlands (2):
  - Het Nederlands Kanker Instituut - Antoni van Leewenhoek Ziekenhuis, Amsterdam
  - Erasmus Medical Center, Rotterdam
- Spain (6):
  - Quiron Salud Barcelona, Barcelona
  - Vall d'Heborn University Hospital - VHIO, Barcelona
  - Clinica Universidad de Navarra, Madrid
  - Quiron Salud Madrid, Madrid
  - Virgen De La Victoria, Málaga
  - Hospital Universitario Virgen De La Macarena, Seville